CLINICAL TRIAL: NCT01379833
Title: Prevalence of Decreased Corneal Sensation in Patients With Chronic Inflammatory Demyelinating Polyneuropathy
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Dent Neurological Institute, Buffalo, NY (Unknown); Fichte, Endl & Elmer Eyecare (Other)
Responsible Party: Principal Investigator, Sangita Patel, Principal Investigator, State University of New York at Buffalo
Other Study IDs: OPT0120511
Record Dates: First submitted 2011-06-16; First posted 2011-06-23 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Chronic Inflammatory Demyelinating Polyneuropathy; Neurotrophic corneal ulcer
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects: Subjects are patients with CIDP
- Controls: Controls are age-matched people without CIDP

SUMMARY:
Chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) is a demyelinating chronic progressive or relapsing neuropathy believed to be secondary to an autoimmune response against peripheral nerve antigens.5 We have observed two patients with CIDP with decreased corneal sensation who also suffered neurotrophic corneal ulcers and severe visual loss in the affected eyes. We want to explore the relationship of CIDP and corneal sensitivity. Our hypothesis is that people with CIDP have decreased corneal sensation compared to those without. We plan to perform a prospective study measuring corneal sensation in patients (proposed n=10) with CIDP and without to determine (1) if a difference exists in patients with CIDP compared to controls and (2) the magnitude of the difference. If a difference is detected in corneal sensitivity in patients with CIDP, this awareness amongst physicians and patients may help prevent blinding complications.

DETAILED DESCRIPTION:
INTRODUCTION The prevalence of CIDP ranges from 0.8 to 8.4 per 100 000.5 This broad range may reflect the use of different diagnostic criteria, as recently confirmed by an epidemiologic study on UK population. Over 50% of the patients may have temporary severe disability during the course of their disease and approximately 10% eventually become persistently disabled or die because of the illness.

CIDP may affect any nerve plexus in the body. However, diagnostic criteria leans towards nerve conduction studies in the limbs and denervation in other organ systems might be overlooked. Sensory innervation of the cornea is provided by the ophthalmic branch of the trigeminal nerve via the anterior ciliary nerves. A relatively small number (50-450) of primary sensory neurons from the ipsilateral trigeminal ganglion send their peripheral axons to the cornea and branch extensively within the corneal tissue. To maintain corneal transparency, all peripheral axons of corneal neurons lose the myelin sheath when they enter the corneal stroma. Fibers spread in a radial fashion parallel to the corneal surface.1

Our proposed study will explore the relationship of decreased corneal sensation, a potentially devastating eye condition secondary to CIDP. Decreased corneal sensation may lead to neurotrophic keratitis; which describes corneal diseases due to impairment or loss of corneal sensation leading to epithelial defects and corneal ulcers. This may be caused by many ocular and systemic diseases such as Diabetes or Stroke. Corneal innervation is important for the maintenance of corneal structure and function, and provides protective mechanisms against factors that might be potentially damaging to the cornea. Innervation also plays an important trophic function in corneal repair in relation to disease, trauma or surgery. Denervation and decreased corneal sensitivity are associated with impairment of epithelial and endothelial cell function, increased epithelial and endothelial permeability, decreased cell migration and cell mitosis. In addition, denervated corneas are predisposed to epithelial or stromal abnormalities, recurrent erosion, impaired wound healing and infection.2

Although corneal nerves lose their myelin sheath as they enter the stroma, the association of a demyelinating disease affecting these nerves cannot be excluded. This may be because trigeminal nerves can be affected at different levels (the nucleus in the pons, the Gasserian ganglion, the trigeminal ophthalmic branch, the nasociliary nerve, or the long ciliary nerve). Also, nerves without central myelin throughout their length can be affected in CIDP. For example, CNVIII has peculiar myelin as it has central myelin for the majority of its length, except for a short distal segment which has peripheral myelin.6 There is one case report correlating findings of hearing loss and vestibular dysfunction for over a 6-year period in patients with CIDP.

OUR STUDY

We plan a prospective clinical trial to compare prevalence of decreased corneal sensation and possible decrease in corneal nerves in patients with CIDP previously diagnosed by clinical features and electrophysiologic data as outlined by the American Academy of Neurology10 as compared to patients without CIDP. Patients will be categorized according to the severity of the disease and duration as per their medical records. Exclusion criteria is aimed at those conditions which may reduce corneal sensation such as previous eye trauma, surgery, contact lens use, eye drop use, or previous viral infections of the eye. A routine complete eye exam will be performed along with additional testing for corneal sensation using a standard method. If significant findings are obtained during initial eye exam, subjects will obtain in-vivo confocal imaging at a second site to image corneal nerve fibers. Published standards for corneal sensitivity as well as corneal nerve fiber density via confocal imaging will be used in statistical analysis.

SIGNIFICANCE OF THIS STUDY

Experimental evidence indicates that impairment of corneal sensory nerves induces pathological changes in the anatomic integrity and function of the cornea, particularly in the epithelium. Loss of corneal sensory innervations leads to a decrease in thickness of the corneal epithelium, intracellular swelling, loss of microvilli and abnormal production of the basal lamina. This may lead to impairment in vitality, metabolism, and mitosis of epithelial cells and, consequently, epithelial breakdown. Persistent epithelial defects may lead to chronic ulceration and eventually to compromise of all ocular surface components with severe visual impairment.

If an association is found between CIDP and decreased corneal sensation, this study will be the first one to demonstrate such an association. An increased awareness among physicians about this association may lead to a more careful eye exam in patients with CIDP and detection of early changes of ocular disease which may be treated earlier so that serious blinding complications can be avoided.

FUTURE STUDIES

If a positive association is found between CIDP and decreased corneal sensation, the latter may be added as a supportive criteria in grading the severity of CIDP. CIDP has many treatment modalities available according to its severity and clinical course. Finding decreased corneal sensation in CIDP patients prospectively may lead to a diagnosis of increased disease severity and patients may benefit from more aggressive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be > 18 years of age. Patients with severe CIDP will be enrolled with age-matched controls without CIDP.

Exclusion Criteria:

* Eye disease (prior or current) other than glasses, Prior eye injury/ trauma, Viral infection (HSV/VZV - prior or current) of eye, Use of contact lenses in last month, Prior eye surgery / laser/lasik, and Use of eye drops other than artificial tears.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with severe CIDP.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Corneal Sensitivity
  The most important variable here is corneal sensitivity in study subjects vs. controls. This is a prospective screen to determine if a difference exists before pursuing larger studies. The endpoint for this investigation will be analysis of 10 patients with CIDP and 10 age-matched controls.

SECONDARY OUTCOMES:
Corneal nerve density
  If there is a difference observed in corneal sensation between subjects and controls, then corneal nerve densities in respective corneas will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Surbhi Bansal, M.D., Principal Investigator — Ross Eye Institute, University at Buffalo; Sangita Patel, M.D. PhD., Study Director — Ross Eye Institute, University at Buffalo; Thomas Elmer, M.D., Study Director — Fichte, Endl & Elmer
Locations (1):
- Dent Neurological Institute, Buffalo, New York, United States

REFERENCES:
- [Background] 1. Bonini S et al. Neurotrophic Keratitis. Contemporary Ophthalmology. 2008. 7(2): 1-8. 2. Grupcheva CH et al. Assessing the sub-basal nerve plexus of the living healthy human cornea by in vivo confocal microscopy. Clinical and Experimental Ophthalmology. 2002, 30: 187-190. 3. Malik RA et al. Corneal confocal microscopy: a non-invasive surrogate of nerve fibre damage and repair in diabetic patients. Diabetologia. 2003. 46: 683-688. 4. Merkies IS et al. Understanding the consequences of chronic inflammatory demyelinating polyradiculoneuropathy from impairments to activity and participation restrictions and reduced quality of life: the ICE study. J Peripher Nerv Syst. 2010 Sep;15(3):208-15. 5. Nobile-Orazio E et al. Chronic inflammatory demyelinating polyradiculoneuropathy and multifocal motor neuropathy: treatment update. Current Opinion in Neurology. 2010; 23: 519-523. 6. Oh SJ. Color Atlas of Nerve Biopsy Pathology. 1st Edition. CRC Press LLC, Boca Raton, Florida. Copyright 2002. 7. Patel DV et al. Contemporary in vivo confocal microscopy of the living human cornea using white light and laser scanning techniques: a major review. Clinical and Experimental Ophthalmology 2007; 35: 71-88. 8. Rajabelly YA et al. Electrophysiological sensory demyelination in typical chronic inflammatory demyelinating polyneuropathy. European Journal of Neurology 2010, 17: 939-944. 9. Van den Bergh PYK et al. European Federation of Neurological Societies/Peripheral Nerve Society Guideline on management of chronic inflammatory demyelinating polyradiculoneuropathy: Report of a joint task force of the European Federation of Neurological Societies and the Peripheral Nerve Society - First Revision. European Journal of Neurology. 2010, 17: 356-363. 10. American Academy of Neurology.
- [Derived] Bansal S, Myneni AA, Mu L, Myers BH, Patel SP. Corneal sensitivity in chronic inflammatory demyelinating polyneuropathy. Cornea. 2014 Jul;33(7):703-6. doi: 10.1097/ICO.0000000000000145. PMID 24858016